CLINICAL TRIAL: NCT05138445
Title: Testing the Effectiveness of Fatigue and Activity Management in Work (FAME-W) Self-management Intervention for Individuals With Inflammatory Arthritis
Brief Title: Effectiveness of Fatigue and Activity Management in Work (FAME-W) for Individuals With Inflammatory Arthritis
Acronym: FAME-W
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: St. James Hospital (Unknown); Tallaght University Hospital (Other); Waterford University Hospital (Unknown)
Responsible Party: Principal Investigator, Deirdre Connolly, Professor Deirdre Connolly, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDublinOT
Record Dates: First submitted 2021-11-02; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Inflammatory Arthritis
Keywords: Work disability; Self-management; Fatigue management; Occupational Therapy
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: FAME-W intervention (Experimental): Four-week self-management education programme
  Interventions: Behavioral: FAME-W self-management intervention
- Arm 2: FAME-W handbook (Active Comparator): Self-guided FAME-W handbook
  Interventions: Behavioral: FAME-W Handbook

INTERVENTIONS:
Behavioral: FAME-W self-management intervention — FAME-W is an occupational therapy led, four-week group based self-management intervention. It focuses on providing people with IA skills and confidence to manage demands of their employment and daily life through education on IA, self-management techniques, managing symptoms of fatigue, pain and stress and managing physical and mental health.
  Arms: Arm 1: FAME-W intervention
Behavioral: FAME-W Handbook — Individuals in this arm receive a self-guided FAME-W handbook containing the same information as that covered in the four week FAME-W program
  Arms: Arm 2: FAME-W handbook

SUMMARY:
Many individuals with Inflammatory Arthritis (IA) experience symptoms of pain and fatigue which interfere with work. Over 50% of people with IA report workplace difficulties resulting in sick leave, absenteeism and reduced productivity. Loss of ability to continue paid employment results in physical, emotional and financial hardship for individuals with IA and has societal and economic implications. Previous research has identified pain and fatigue as dominant symptoms that interfere with work capacity and therefore interventions are required to reduce the impact of these symptoms on work activities. The purpose of this study therefore is to test the effectiveness of a 4-week Fatigue and Activity Management Education for Work intervention. The study will use a mixed methods design. A randomized control trial will test the effectiveness of the intervention and a qualitative process evaluation with explore acceptability and participants' experiences of the intervention. Individuals with IA, of working age, will be recruited in Rheumatology outpatient departments of three hospitals. Study participants will be randomly assigned to a four-week online self-management intervention or a self-guided symptom management workbook. Study measures consist of self-report questionnaires related to work and symptom management. All participants will also be invited to an interview to discuss their experience of participating in the study.

DETAILED DESCRIPTION:
Rheumatic diseases (RD) include over 100 different types of arthritis, the most frequently occurring being Rheumatoid Arthritis, Osteoarthritis, Scleroderma, Systemic Lupus erythmatosus and ankylsoing Spondylitis. However, Inflammatory Arthritis (IA) are one of the most common causes of work disability and despite improvements in medical management of IA, up to 50% of people with IA report workplace difficulties resulting in sick leave, absenteeism and reduced productivity.

This study builds on existing research investigating the impact of IA on work performance of individuals. These earlier studies examined how symptoms of fatigue, pain and stress impact on work capacity of individuals with IA. Based on the findings of these studies a self-management program, FAtigue Management Education for Work (FAME-W) was designed to reduce the impact of fatigue, pain and stress on work performance of individuals with IA. Pilot testing of FAME-W, with a non-experimental design, showed improvements in fatigue, work performance, pain and mood following participation in FAME-W. The proposed study will build on this research by testing the effectiveness of FAME-W as a work-focused self-management intervention to increase work performance of individuals with IA.

Project Design and Methodology

Study Aim

The purpose of this study is to test the effectiveness and acceptability of FAME-W to manage the physical, mental and social demands of work of individuals with IA.

Study Objectives

* To test the effectiveness of FAME-W in reducing the impact of fatigue, pain and stress on work performance of individuals with Inflammatory Arthritis.
* To test the effectiveness of FAME-W in improving work ability of individuals with Inflammatory Arthritis
* To explore the acceptability of FAME-W as a work-based self-management intervention for individuals with Inflammatory Arthritis

Study Design

The study methodology will follow the United Kingdom Medical Research Council (MRC) framework for evaluating complex interventions. A complex intervention consists of a number of interacting components such as those included in the FAME-W intervention. The MRC framework recommends collecting quantitative and qualitative data when evaluating complex interventions. This study will therefore use a sequential exploratory mixed methods design.

The quantitative phase will be a pragmatic randomized control trial (RCT) to test the effectiveness of FAME-W as a work focused self-management intervention to improve individuals' ability to manage their work demands. The CONSORT guidelines for the design and reporting of RCTs will be used at all stages from recruitment, randomization, data collection, analysis and reporting. For the purposes of the proposed study, participants will be randomly allocated to either the group based FAME-W intervention or to a handbook only group. Participants randomized to the group-based FAME-W group will attend an online four-week FAME-W program. The participants in handbook only group will be given a self-guided FAME-W handbook.

The qualitative phase will use a Qualitative Descriptive (QD) design to explore participants' experiences and acceptability of FAME-W. QD is frequently used in health research to evaluate the acceptability and sustainability of health-related interventions. It is considered an appropriate methodology for needs assessments and for informing the planning and delivery of clinical interventions.

Sample Size

Based on the previous studies the individual scores for Work Role Functioning (WRF) questionnaire this study is powered for an effect size of 0.7. To detect an 0.7, 100 participants are required (50 for the group intervention and 50 for handbook only group) to show significance at 5% level, 80% power. Participants will be recruited in groups of 12-14 and then allocated to the intervention or control group using random allocation software.

Data collection methods

Quantitative Data:

Patient Reported Outcome Measures (PROMS, outlined below) will be used to collect quantitative data

Qualitative phase: Qualitative data will be collected from individual interviews and focus groups.

Data collection will be carried out immediately before FAME-W commences, immediately following completion of FAME-W, and 3 months following completion of the program.

Data analysis Quantitative data: Baseline characteristics will be analyzed using descriptive statistics. Multilevel linear regression will be used to examine differences between groups for the primary and secondary outcome measures. Statistical significance at p<0.05 will be assumed throughout.

Qualitative data: Semi-structured interviews will be audio-taped and transcribed. Data analysis will be guided by Braun and Clarke's seven stage thematic analysis of qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Inflammatory Arthritis,
* In full-time or part-time employment
* Must be able to provide informed consent,
* Must be able to participate in a four-week group-based self-management intervention
* Must have access to an electronic device and stable internet access

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Work Role Functioning Questionnaire | Three months
  Work Role Functioning questionnaire is a 27-self-report questionnaire that measures an individual's ability to meet demands of five categories of work: scheduling, output, psychical, mental and social demands. All 27 items are scored on a five point scale, with a score of four given for the response 'difficult none of the time' and a score of zero representing 'difficult all of the time'. Each of the five sub-scales are scored separately. A score is established by adding the response of each item, calculating the average and multiplying this by 25 to achieve an overall percentage. The overall percent can range from 0% (difficult all of the time), to 100% (never difficult) meeting the demands of the job.

SECONDARY OUTCOMES:
Euro QoL 5 Dimensions -5 levels (5D-5L) | Three months
  Euro QoL 5 Dimensions -5 levels scale evaluates the health-related quality of life and compromises two components: a health descriptive component and a visual analog scale (VAS) . It has five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each category is scored from 1 (no problem) to 5 (extreme problems). Scores range from 1-25. Higher scores represent higher levels of difficulty. A visual analogue scale measures self-perception of health-related quality of life on a scale of 0-100. Higher scores represent better levels of health-related quality of life.
Multidimensional Fatigue Inventory | Three months
  Multidimensional Fatigue Inventory evaluates five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. It is a 20-item self-report questionnaire scored from 4 to 20. Higher scores indicate higher levels of fatigue
Arthritis Work Spillover | Three months
  Arthritis Work Spillover is designed to assess the extent to which the demands of arthritis interfere with work performance and the extent to which work interferes with managing arthritis. Items are scored on a 5-point Likert scale where 1= strongly disagree and 5 = strongly agree. Scores range from 6 - 30. Higher scores indicate higher level of interference between work and arthritis
Hospital Anxiety and Depression scale (HADS) | Three months
  This scale is a self-report measure with two sub scales for measuring anxiety and depression. Each scale contains seven items and ranges from a score of 0 to 21. Higher scores indicate higher levels of anxiety and depression.
The Stanford Arthritis Self-Efficacy Scale Short Form | Three months
  The Stanford Arthritis Self-Efficacy Scale Short Form is a self-administered, 20-item disease-specific questionnaire suitable for all types of arthritis. It consists of three sub scales: physical function, other symptoms, and pain.Each item is scored between one (very uncertain) and 10 (very certain) with higher scores indicating higher levels of self-efficacy.
The Arthritis Impact Measurement Scale | Three months
  The Arthritis Impact Measurement Scale was developed to measure the physical, mental, and emotional well-being of individuals with arthritis. It consists of five domains: physical functioning, symptoms, mood/affect, social interaction, and work-role components. Scores range from 0-10. Higher scores indicate poorer overall health.
The Short Form McGill Pain Questionnaire | Three months
  The Short Form McGill Pain Questionnaire was developed to measure pain in adults with chronic pain, including individuals with rheumatic conditions. Scores range from zero to 10 with higher scores indicating higher levels of pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Connolly, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Trinity College Dublin, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data may be shared for results presented in publications of quantitative data on request to the study contact person.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for six months following related publications
Access Criteria: Requests for data sharing can be made to the study central contact person via email.

REFERENCES:
- [Derived] Karkon S, Bennett KE, O'Shea F, Doran M, Connolly D. Testing the effectiveness of a Fatigue and Activity Management Education for Work (FAME-W) intervention for individuals with inflammatory arthritis: Study protocol for a randomized control trial. Musculoskeletal Care. 2023 Dec;21(4):1629-1638. doi: 10.1002/msc.1839. Epub 2023 Nov 7. PMID 37937322